CLINICAL TRIAL: NCT05871801
Title: Comparative Study of Predictive Models of Inadequate Colonic Preparation
Brief Title: Predictive Models of Inadequate Colonic Preparation
Acronym: Quality
Status: Completed | Type: Observational
Sponsor: Manuel Hernandez-Guerra, MD (Other)
Responsible Party: Sponsor-Investigator, Manuel Hernandez-Guerra, MD, Clinical Professor, University of La Laguna
Organization: University of La Laguna (Other)
Other Study IDs: CHUC_2022_87
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cleansing Quality of the Colon
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bowel preparation for colonoscopy — one day liquid diet will be administered to every patient included in the study and: split-dose bowel preparation with 4 Liters of Polyethylenglycol (PEG) solution, 2 Liters of PEG-Asccorbic acid or 2L sodium picosulphate.
Device: Colonoscopic examination — Colonoscopy will be performed to every patient included in the study

SUMMARY:
The main purpose of the study is to evaluate in a prospective cohort of patients with an appointment for the performance of an outpatient colonoscopy the prediction of the quality of colonic cleansing through the use of 3 predictive models.

The colon cleansing quality will be assessed by a validated scale (Boston Bowel Preparation Scale, BBPS). Patients will be prepared with polyethylene glycol (PEG), PEG plus ascorbic acid (PEG-Asc) or sodium picosulfate-oxide magnesium solution (PS).

DETAILED DESCRIPTION:
Although, current guidelines recommend a rate of inadequate bowel cleansing for colonoscopy not higher than 10-15%, in clinical practice poor bowel cleansing in endoscopy units ranged between 6.8% and 33%. The determinants of poor cleanliness have been evaluated in different studies and can be classified into patient-dependent predictors, which include demographic, socioeconomic and clinical variables, variables dependent on the preparation protocol, including the assigned diet, the type of preparation, its fractionation and the space of time elapsed between the last intake and the colonoscopy, and the tolerance mainly attributed to the volume and taste of the evacuating preparation The American Association of Gastrointestinal Endoscopy recommends the administration of additional preparation to these patients with a higher probability of inadequate preparation. Once non-compliance and lack of tolerance to cleaning protocols are excluded, the reason for inadequate preparation is usually the lack of effectiveness of the cleaning protocol. Therefore, it is advisable to select patients who can benefit from supplemented cleaning preparation or intensified cleaning protocols.

There are so far 4 published predictive models that incorporate clinical variables with the aim of determining patients who are candidates for intensified preparations. Of the models mentioned in the previous studies, only 3 are clearly detailed in the corresponding articles.

The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information.

Subsequently, the colonoscopy will be performed and the cleaning quality will be scored according to the BBPS considering suboptimal a cleaning quality of less than 2 points in a segment of the colon.

The bowel cleansing quality following BBPS will be assessed by the endoscopist

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* To sign the informed consent,
* Patients with indication of outpatient colonoscopy
* Patients ingesting preparation

Exclusion Criteria:

* Resection of more than one colon segment.
* Ileus, intestinal obstruction, megacolon.
* Poorly controlled hypertension (HTAS> 180 HTAD> 100).
* Terminal renal failure (pre-dialysis or dialysis).
* Congestive heart failure (NYHA III-IV).
* Acute liver failure.
* Severe psychiatric illness.
* Dementia with difficulty in the intake of the preparation.
* Pregnancy or breastfeeding.
* Refusal to participate in the study.
* Allergies.
* Incomplete colonoscopy except for poor bowel cleansing

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The researchers will offer to participate in the study to outpatients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of poor bowel cleansing assessed by the Boston Bowel Preparation Scale | 3 months
  Quality of bowel cleansing assessed by the Boston Bowel Preparation Scale. This scale goes from 0 (no preparation) to 3 points (excellent preparation) in the three segments of the colon (proximal, transverse and distal). The maximum score is 9 points

SECONDARY OUTCOMES:
Number of predictive factors of poor bowel cleansing | 3 months
  To evaluate the factors associated with inadequate colonic cleaning in this cohort of patients with the aim of improving the models described above

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno García, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No
Data will no be available to other researchers

REFERENCES:
- [Background] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Background] Berger A, Cesbron-Metivier E, Bertrais S, Olivier A, Becq A, Boursier J, Lannes A, Luet D, Pateu E, Dib N, Caroli-Bosc FX, Vitellius C, Cales P. A predictive score of inadequate bowel preparation based on a self-administered questionnaire: PREPA-CO. Clin Res Hepatol Gastroenterol. 2021 Jul;45(4):101693. doi: 10.1016/j.clinre.2021.101693. Epub 2021 Apr 20. PMID 33852957
- [Background] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690